CLINICAL TRIAL: NCT01754220
Title: The Effects of Alvokast (Montelukast) in Patients With Chronic Cough
Brief Title: Open-label Study of the Effects of Montelukast in Patients With Chronic Cough
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association Asthma, Bulgaria (Other)
Responsible Party: Principal Investigator, Prof. Todor Popov, Professor, Association Asthma, Bulgaria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALKA-03-12
Record Dates: First submitted 2012-11-03; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Coughing
MeSH Terms: conditions — Cough | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Montelukast (Active Comparator): Montelukast tablets: adults - 10 mg, children - 5mg taken daily for two weeks
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Montelukast is a leukotriene receptor antagonist
  Other Names: Alvokast

SUMMARY:
Montelukast, a leukotriene receptor antagonist, is likely to be effective in the treatment of chronic cough and this could be made objective by measuring cough threshold before and after two weeks of treatment.

DETAILED DESCRIPTION:
Chronic cough is typically defined as cough that persists for longer than 8 weeks and is the most common presenting symptom in adults who seek medical treatment in an ambulatory setting. Prospective studies have shown that three conditions account for the etiologic cause of chronic cough in the largest part of immunocompetent, nonsmoking patients with normal chest radiograph findings. In order of frequency, they are upper airway cough syndrome (UACS), previously referred to as postnasal drip syndrome (PNDS), asthma and gastroesophageal reflux disease (GERD). UACS comprises many different conditions including PNDS, acute sinusitis, allergic rhinitis, non-allergic rhinitis (postinfectious rhinitis, rhinitis medicamentosa, vasomotor rhinitis, rhinitis due to physical or chemical irritants). Cough occurs in all asthmatics, and in a subset of patients with cough-variant asthma (CVA), it is the only presenting symptom. In these cases it is well controlled with inhaled corticosteroids and beta-2 agonists. GERD is another cause that should be contemplated when anti-tussive or anti-inflammatory/anti-allergic treatment do not render results and when there are presenting symptoms suggestive of it. Moreover, factors like smoking and use of ACE-inhibitors should also be taken into account.

Leukotrienes are very important agents in the inflammatory response. It is known that they are contributing significantly to the pathological processes in asthma. Montelukast is a leukotriene receptor antagonist which blocks the bonding of leukotrienes to their receptors thus inhibiting their inflammatory, bronchoconstrictive and mucosecretory effects. Multiple clinical trials have demonstrated the ability of the leukotriene antagonists to improve symptoms, pulmonary function and bronchial hyperresponsiveness in patients with asthma. However, not much is known about their effects in people with chronic cough. Studies have been carried out in an attempt to find out the effects of montelukast in some forms of chronic cough. Nevertheless, the impact of montelukast on objective parameters such as cough reflex threshold, has not been explored. The investigators also reckon that montelukast will affect exhaled breath temperature - a novel surrogate marker of airway inflammation recognized lately

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic cough: cough persisting for more than 8 consecutive weeks

Exclusion Criteria:

* Current use of ACE-inhibitors
* Use of systemic steroids in the last 4 weeks
* COPD
* Pregnancy
* Concomitant severe disease
* Smoking

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in the cough reflex parameters (C2 and C5) before and after two weeks of treatment with montelukast | 7 months
Difference in average scores on modified Leicester Cough Questionnaire (LCQ) before and after two weeks of treatment with montelukast | 7 months

SECONDARY OUTCOMES:
Difference in pulmonary function parameters (FVC, FEV1, PEF), before and after two weeks of treatment with montelukast | 7 months
Difference in Exhaled breath temperature (EBT) before and after two weeks of treatment with montelukast | 7 months
Difference in laboratory markers (CBC, CRP, total IgE, ESP, MPO) before and after two weeks of treatment with montelukast | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Todor A Popov, MD, Phd, Principal Investigator — Association Asthma, Bulgaria
Locations (1):
- Clinic of Allergy and Asthma, University Hospital "Alexandrovska", Sofia, Sofia, Bulgaria

REFERENCES:
- [Background] Palombini BC, Villanova CA, Araujo E, Gastal OL, Alt DC, Stolz DP, Palombini CO. A pathogenic triad in chronic cough: asthma, postnasal drip syndrome, and gastroesophageal reflux disease. Chest. 1999 Aug;116(2):279-84. doi: 10.1378/chest.116.2.279. PMID 10453852
- [Background] Paredi P, Caramori G, Cramer D, Ward S, Ciaccia A, Papi A, Kharitonov SA, Barnes PJ. Slower rise of exhaled breath temperature in chronic obstructive pulmonary disease. Eur Respir J. 2003 Mar;21(3):439-43. doi: 10.1183/09031936.03.00061902. PMID 12661998
- [Derived] Mincheva RK, Kralimarkova TZ, Rasheva M, Dimitrov Z, Nedeva D, Staevska M, Papochieva V, Perenovska P, Bacheva K, Dimitrov VD, Popov TA. A real - life observational pilot study to evaluate the effects of two-week treatment with montelukast in patients with chronic cough. Cough. 2014 Mar 20;10(1):2. doi: 10.1186/1745-9974-10-2. PMID 24649919